CLINICAL TRIAL: NCT07270237
Title: Development and Evaluation of Ultrasound Imaging Acquisition and Analysis Methods
Brief Title: A Study of Multiparametric Ultrasound Imaging Methods
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 25-299
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Pancreatic Cancer; Thyroid Nodule
Keywords: Ultrasound; mpUS; 25-299
MeSH Terms: conditions — Pancreatic Neoplasms; Thyroid Nodule | interventions — Diagnostic Imaging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Multiparametric endoscopic (mpEUS) imaging of patients at high-risk for pancreatic cancer (Experimental): Subjects will undergo add-on mpEUS imaging during their standard of care EUS imaging and will add up to approximately 15 minutes of added scan time.
  Interventions: Diagnostic Test: Multiparametric ultrasound (mpUS) imaging
- Multiparametric endoscopic (mpEUS) imaging of patients with pancreatic ductal adenocarcinoma (Experimental): Subjects will undergo add-on mpEUS imaging during their standard EUS procedure and will add up to approximately 15 minutes of added scan time.
  Interventions: Diagnostic Test: Multiparametric ultrasound (mpUS) imaging
- Thyroid nodule assessment with multiparametric ultrasound (mpUS) imaging (Experimental): Subjects will undergo add-on mpUS imaging at the beginning of their standard of care ultrasound procedure and will add up to approximately 5 minutes of added scan time.
  Interventions: Diagnostic Test: Multiparametric ultrasound (mpUS) imaging

INTERVENTIONS:
Diagnostic Test: Multiparametric ultrasound (mpUS) imaging — Patients will undergo the added research sequences at any point during their standard of care ultrasound scans, adding up to approximately 15 minutes of added scan time. The only non-routine measurements will be the research ultrasound data.

SUMMARY:
The researchers are doing this study to see how well a type of ultrasound imaging called multiparametric ultrasound (mpUS), can be used to examine, evaluate, and provide information about different cancerous and non-cancerous tissue. The researchers will compare the results of mpUS imaging to standard ultrasound imaging and other standard tests.

mpUS imaging is a type of ultrasound imaging that combines different ultrasound methods and analysis to create a more detailed and accurate assessment of tissue. Standard ultrasound provides a basic image of tissue structure, but mpUS imaging can also show blood vessels, blood flow, and detailed tissue structure (microstructure). The researchers think that mpUS may be a better way for evaluating cancer because it combines different ultrasound methods to assess tissue.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1 - Feasibility of multiparametric endoscopic ultrasound (mpEUS) imaging of patients at high-risk for pancreatic cancer:

Patient Group: those having standard endoscopic ultrasounds because they are at high risk of pancreatic cancer Participants enrolled into the Memorial Sloan Kettering Cancer Center Pancreatic Registry protocol (IRB#: 02-102) will be eligible for this study. Specifically, related individuals without pancreatic cancer who are at-risk for developing pancreatic cancer and meet all of the following criteria (family health history will be self-reported):

* 10 years younger than the earliest pancreatic cancer diagnosis in the family
* Be at least 50 years old
* Be at least 40 years old if diagnosed with FAMMM syndrome (CDKN2A/p16) or Hereditary Pancreatitis (PRSS1, SPINK1/PST1, CTRC, CPA1 or other candidate hereditary pancreatitis genes)
* Be at least 35 years old if diagnosed with Peutz-Jeghers syndrome (STK11 aka LKB1)
* Not pregnant and not Nursing
* Relatives at least 21 years old with other high-risk clinical criteria that warrants pancreatic cancer surveillance or follow-up as determined by the project leader (Dr. Vineet Rolston)
* Must agree to be contacted for follow-up
* Must satisfy at least one of the following 4 criteria:

  1. Have at least two affected relatives who are a first-degree relative to each other, of whom at least one is a first degree relative to the individual OR have at least two affected first-degree relatives on the same side of the family.
  2. Have at least one first- or second-degree affected relative and have germline genetic test results that confirm a likely pathogenic or pathogenic variant in at least one of the following genes:

     1. APC (Familial Adenomatous Polyposis (FAP) and Attenuated FAP syndrome
     2. BRCA1(Hereditary Breast and Ovarian Cancer Symptoms)
     3. MLH1, MSH2, MSH6, PMS2, or EPCAM (Lynch Syndrome)
     4. PALB2
     5. TP53 (Li-Fraumeni Syndrome)
     6. Other established pancreatic cancer predisposition gene per project leader's discretion
  3. Have germline genetic test results that confirm a likely pathogenic or pathogenic variant in one or more of the following genes:

     1. CDKN2A/p16 (Familial Atypical Multiple Mole Melanoma Syndrome (FAMMM))
     2. STK11 aka LKB1 (Peutz-Jeghers Syndrome)
     3. PRSS1, SPINK1/PST1, CTRC, CPA1 or other candidate hereditary pancreatitis genes per project leader's discretion
     4. ATM (ataxia telangiectasia mutated)
     5. BRCA 2(Hereditary Breast and Ovarian Cancer Symptoms)
  4. Relatives at least 21 years old with other high-risk clinical criteria that warrants pancreatic cancer surveillance or follow-up as determined the project leader (Dr. Vineet Rolston)

Cohort 2 - Multiparametric endoscopic ultrasound imaging (mpEUS) of patients with pancreatic ductal adenocarcinoma:

Patient Group: those with pancreatic cancer having endoscopic ultrasound-guided biopsies

Patients will be entered into the study if they meet the following criteria:

* Patients with pancreatic ductal adenocarcinoma
* Are undergoing endoscopic ultrasound-guided tissue core biopsy as part of their standard of care
* Not pregnant and not nursing

Cohort 3 - Thyroid nodule assessment with multiparametric ultrasound (mpUS) imaging:

Patient Group: those with a thyroid nodule that will be biopsied whether they have known cancer or not

* Are undergoing ultrasound-guided thyroid biopsy as part of their standard of care
* Not pregnant and not nursing

Healthy Volunteers will be entered into the study if they meet the following criteria:

* No known cancer diagnosis or thyroid nodules
* Age ≥ 18
* Able to understand and give informed consent
* Not pregnant and not nursing

Exclusion Criteria:

Cohort 2 - Multiparametric endoscopic ultrasound imaging (mpEUS) of patients with pancreatic ductal adenocarcinoma:

* Unable to sign an informed consent for medical or other reasons; residents outside the continental United States
* Under 18 years of age

Cohort 3 -Thyroid nodule assessment with multiparametric ultrasound (mpUS) imaging

* Unable to sign an informed consent for medical or other reasons; residents outside the continental United States
* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
investigate the feasibility of mpEUS imaging | 1 day
  the feasibility rate will be estimated and reported using the corresponding sample proportion, along with exact binomial 95% confidence intervals. The mpEUS technique will be considered feasible if it is able to visualize/quantify parameters in at least 21 patients out of the 30 patients.

CONTACTS AND LOCATIONS:
Overall Officials: Mark T Burgess, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Consent Only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent Only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent Only), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent Only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Consent Only), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/